CLINICAL TRIAL: NCT04430712
Title: Immune Checkpoint Inhibitors and Atherosclerotic Plaque Volume in Patients With Non-Small Cell Lung Cancer: A Case-Control Study
Brief Title: Immune Checkpoint Inhibitors and Atherosclerotic Plaque Volume
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Tomas G. Neilan, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2020P000361
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; Immune Checkpoint Inhibitor; Atherosclerosis
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, investigators plan to test whether Immune Checkpoint Inhibitor (ICI) treatment leads to an accelerated progression of atherosclerosis in patients with lung cancer. Atherosclerosis is an immune-mediated inflammatory disease and these same checkpoints being targeted for cancer are critical negative regulators of atherosclerosis in animal and cellular models. Aortic plaque progression will be compared between cases (on ICI) and controls from pre-ICI to post-ICI among patients with non-small cell lung cancer. Groups will be matched for age, cancer type and stage and cardiovascular risk factors. Traditional markers of cardiovascular (CVD) risk and cancer-specific factors (ICI mono- and combination therapy, number of cycles, occurrence of immune-related adverse events, chest radiation, steroid use) will be associated with the change in aortic plaque volume.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* Subjects with non-small cell lung cancer treated with Immune Checkpoint Inhibitors.
* Available contrast enhanced CT scans of the chest both immediately pre-ICI (< 1 month) and latest follow-up.

Controls:

* Subjects with non-small cell lung cancer, age, cancer stage and cardiovascular risk factor matched to cases.
* Available contrast enhanced CT scan of the chest at two time-points at a similar interval between scans as the cases.

Exclusion Criteria:

none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-small cell lung cancer from a single tertiary care center in the United States.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-08-12 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Change in aortic plaque volume | Three years
  The change of plaque burden after starting ICIs will be calculated and compared with the pre-ICI study. The change in plaque burden in controls will be calculated and compared from two studies at a similar median interval as ICI cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Drobni ZD, Gongora C, Taron J, Suero-Abreu GA, Karady J, Gilman HK, Supraja S, Nikolaidou S, Leeper N, Merkely B, Maurovich-Horvat P, Foldyna B, Neilan TG. Impact of immune checkpoint inhibitors on atherosclerosis progression in patients with lung cancer. J Immunother Cancer. 2023 Jul;11(7):e007307. doi: 10.1136/jitc-2023-007307. PMID 37433718